CLINICAL TRIAL: NCT04936425
Title: Comparison of Stent Suturing Versus OTSC Stentfix in Preventing Esophageal Stent Migration in Non-Stricture Esophageal Lesions
Brief Title: Comparison of Stent Suturing Versus OTSC Stentfix
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-01140
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Stent Fixation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded as to which study arm they are in, in order to avoid any bias they may have.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- OTSC Stentfix (Experimental)
  Interventions: Device: OTSC Stentfix
- Stent Suturing (No Intervention)

INTERVENTIONS:
Device: OTSC Stentfix — The OTSC stentfix will be placed during upper endoscopy after a self-expanding metal stent has been deployed.
  Arms: OTSC Stentfix

SUMMARY:
The purpose of this study is to investigate whether OTSC stentfix is a feasible, safe, and efficient device that can be used for esophageal stent fixation (to prevent stent migration) in patients with benign, non-stricture esophageal lesions, including leaks, perforation, and fistulae. Currently, self-expandable metal stents (SEMS) have a risk of migration which can lead to adverse events such as bleeding and perforation. There has been clinical experience demonstrating that stent suturing can prevent stent migration. However, stent suturing can significantly increase endoscopic procedural time. The use of OTSC stentfix for stent fixation is promising as it is likely less time-consuming and less technically difficult, with likely a similar rate of fixation and migration. This non-inferiority study aims to investigate how OTSC stentfix functions as compared to stent suturing. If OTSC stentfix is at least comparable to stent suturing, it can reduce endoscopy procedural times, minimize peri-endoscopic risks, and minimize adverse events related to stent migration.

ELIGIBILITY:
Inclusion Criteria:

* All adults (18+ years)
* Have benign, non-stricture esophageal lesions (i.e. fistulae, perforation, leaks) warranting esophageal stent placement as an inpatient or outpatient
* Ability to consent to stent fixation.

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-21 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Average rate of stent migration | 48 weeks

SECONDARY OUTCOMES:
Procedural time needed for stent fixation | 120 minutes
Duration of time until stent migration for stents that fail fixation | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Haber, MD, Principal Investigator — NYU Langone Health; Lauren Khanna, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be share upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to sofia.yuen@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.